CLINICAL TRIAL: NCT06074081
Title: Comparison of 4-weeks of Motor Relearning Program and Mirror Therapy in Improving Upper Limb Motor Function in Stroke Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yusra Medical and Dental College (Other)
Responsible Party: Principal Investigator, Maham Nasir, Head of Physical Therapy Department, Yusra Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Motor Relearning Program
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Stroke
Keywords: Motor Relearning Program; Mirror therapy
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Participants are divided into 2 groups Patients in experimental group will receive treatment through Motor-relearning program. Patient in controlled group will receive treatment through mirror therapy .
Who Masked: Participant
Masking Description: It is a single blinded study in which participants will be allocated into 2 groups by using coin flip method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor relearning program (Experimental): Patients in this group will receive treatment through Motor-relearning programme. Patients will be instructed to perform multiple task like holding object, elbow extension/flexion and multiple movements of shoulder joint. This group will receive MRP for about time duration of 4 weeks,3 days per week,2 hours session per day.
  Interventions: Other: motor relearning program
- mirror therapy (Other): Patient in this group will receive treatment through mirror therapy. Patient will sit in such a way that the mirror will be placed in perpendicular direction on a table. Sound limb will place in front of mirror and affected limb will place behind the mirror. Patient will receive visual feedback from sound limb. This group will receive MT for about 4 weeks, 3 days per week, 2 hours session per day.
  Interventions: Other: mirror therapy

INTERVENTIONS:
Other: motor relearning program — MRP is a therapy to regain particular motor function and neglecting accessory movements by engaging cognitive behavior .
  Arms: motor relearning program
Other: mirror therapy — Mirror therapy enhance functional activities in patient with hemiplegic stroke. For betterment of result high quality methodological studies and larger sample size is required.
  Arms: mirror therapy

SUMMARY:
Cerebrovascular accident(CVA) or stroke is one of common condition affecting people in developed and underdeveloped countries.

MRP is a therapy to regain particular motor function and neglecting accessory movements by engaging cognitive behavior.

Mirror therapy enhance functional activities in patient with hemiplegic stroke. For betterment of result high quality methodological studies and larger sample size is required.

DETAILED DESCRIPTION:
Cerebrovascular accident(CVA) or stroke is one of common condition affecting people in developed and underdeveloped countries. Mostly patient with stroke face many disabilities and the most important one is upper limb motor impairment. For the optimization of upper extremity and prevention of patient from permanent disability it is essential to promotes Neuro-rehabilitation interventions. Physiotherapy techniques need to be monotonous, thorough and task oriented for neuroplasticity to generate better recovery. There is notable enhancement in ADLS when the rehabilitation program starts within 16 hours to 6 months after stroke In improving upper extremity motor functions there are tremendous types of techniques used i.e. Proprioceptive neuromuscular facilitation(PNF),Brunnstorm, Bobath therapy, Motor relearning program(MRP),Constraint induced movement therapy(CIMT) and Mirror therapy(MT).Out of which we are using two basic techniques i.e. motor relearning program(MRP) and mirror therapy(MT).Mirror therapy enhance functional activities in patient with hemiplegic stroke. For betterment of result high quality methodological studies and larger sample size is required. Mirror therapy enhance functional activities in patient with hemiplegic stroke. MRP is a therapy to regain particular motor function and neglecting accessory movements by engaging cognitive behavior .MRP is a therapy to regain particular motor function and neglecting accessory movements by engaging cognitive behavior.

ELIGIBILITY:
Inclusion Criteria

* Acute(hemiplegic attack within 1-2 weeks) and sub-acute stroke(hemiplegic attack within 3- 11 weeks).
* 20 to 80 years.
* No physical deformity prior to stroke
* No history of serious underlying pathology and structural deformities.

Exclusion Criteria:

* Patient with chronic hemiplegic stroke.
* Patient with congenital deformity.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
fugl meyer assessment scale (FMA) | upto 4 weeks
  This test is recommended for checking functional return of patient having impairments with stroke.Test consists on the base of assessing patient with moving limb in low tone movements or synergistic pattern and then move actively back to normal function. Total scoring for upper limb is 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Maham Nasir, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jan S, Arsh A, Darain H, Gul S. A randomized control trial comparing the effects of motor relearning programme and mirror therapy for improving upper limb motor functions in stroke patients. J Pak Med Assoc. 2019 Sep;69(9):1242-1245. PMID 31511706
- [Background] Ng JC, Churojana A, Pongpech S, Vu LD, Sadikin C, Mahadevan J, Subramaniam J, Jocson VE, Lee W. Current state of acute stroke care in Southeast Asian countries. Interv Neuroradiol. 2019 Jun;25(3):291-296. doi: 10.1177/1591019918811804. Epub 2018 Nov 21. PMID 30463501
- [Background] Zhang Y, Xing Y, Li C, Hua Y, Hu J, Wang Y, Ya R, Meng Q, Bai Y. Mirror therapy for unilateral neglect after stroke: A systematic review. Eur J Neurol. 2022 Jan;29(1):358-371. doi: 10.1111/ene.15122. Epub 2021 Oct 5. PMID 34558762
- [Background] Ullah I, Arsh A, Zahir A, Jan S. Motor relearning program along with electrical stimulation for improving upper limb function in stroke patients: A quasi experimental study. Pak J Med Sci. 2020 Nov-Dec;36(7):1613-1617. doi: 10.12669/pjms.36.7.2351. PMID 33235584
- [Background] Gandhi DB, Sterba A, Khatter H, Pandian JD. Mirror Therapy in Stroke Rehabilitation: Current Perspectives. Ther Clin Risk Manag. 2020 Feb 7;16:75-85. doi: 10.2147/TCRM.S206883. eCollection 2020. PMID 32103968
- [Background] improved upper limb motor recovery and level of independence after stroke: a randomized controlled trial. CadernosBrasileiros de TerapiaOcupacional. 2022 Sep 2;30.
- [Background] Zeng W, Guo Y, Wu G, Liu X, Fang Q. Mirror therapy for motor function of the upper extremity in patients with stroke: A meta-analysis. J Rehabil Med. 2018 Jan 10;50(1):8-15. doi: 10.2340/16501977-2287. PMID 29077129
- [Background] Hsieh YW, Lin YH, Zhu JD, Wu CY, Lin YP, Chen CC. Treatment Effects of Upper Limb Action Observation Therapy and Mirror Therapy on Rehabilitation Outcomes after Subacute Stroke: A Pilot Study. Behav Neurol. 2020 Jan 2;2020:6250524. doi: 10.1155/2020/6250524. eCollection 2020. PMID 32377266
- [Background] Maratis J, Wahidin A, Ivanali K. COMPARE THE EFFECTIVENESS OF CONSTRAINT INDUCED MOVEMENT THERAPY AND MOTOR RELEARNING PROGRAMME IN POST STROKE PATIENTS. In Academic Physiotherapy Conference Proceeding 2021 (pp. 179-190).
- [Background] Rehme AK, Eickhoff SB, Rottschy C, Fink GR, Grefkes C. Activation likelihood estimation meta-analysis of motor-related neural activity after stroke. Neuroimage. 2012 Feb 1;59(3):2771-82. doi: 10.1016/j.neuroimage.2011.10.023. Epub 2011 Oct 17. PMID 22023742
- [Background] Hassani Z, Mokhtarinia HR, Kahlaee AH, Gabel CP. Translation, Validity, and Reliability of the Upper Extremity Fugl-Meyer Assessment (FMA-UE) in Persian Speaking Stroke Patients. Iranian Rehabilitation Journal. 2022 Mar 10;20:37-46.
- [Background] Malouin F, Pichard L, Bonneau C, Durand A, Corriveau D. Evaluating motor recovery early after stroke: comparison of the Fugl-Meyer Assessment and the Motor Assessment Scale. Arch Phys Med Rehabil. 1994 Nov;75(11):1206-12. doi: 10.1016/0003-9993(94)90006-x. PMID 7979930
- [Background] Platz T, Pinkowski C, van Wijck F, Kim IH, di Bella P, Johnson G. Reliability and validity of arm function assessment with standardized guidelines for the Fugl-Meyer Test, Action Research Arm Test and Box and Block Test: a multicentre study. Clin Rehabil. 2005 Jun;19(4):404-11. doi: 10.1191/0269215505cr832oa. PMID 15929509
- [Background] Arfianti L, Rochman F, Hidayati HB, Subadi I. The addition of mirror therapy
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Fagundes NCF, Almeida APCPSC, Vilhena KFB, Magno MB, Maia LC, Lima RR. Periodontitis As A Risk Factor For Stroke: A Systematic Review And Meta-Analysis. Vasc Health Risk Manag. 2019 Nov 6;15:519-532. doi: 10.2147/VHRM.S204097. eCollection 2019. PMID 31806984